CLINICAL TRIAL: NCT04650789
Title: Longitudinal Study of Frailty in Shanghai Older People
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: Shanghai Frailty Survey
Record Dates: First submitted 2020-08-24; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-05

CONDITIONS: Frailty
Keywords: Frailty; Longitudinal cohort study; prevalence
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the prevalence of Frailty in community older residents.

DETAILED DESCRIPTION:
Detailed Description:

1. Objective:

   * To investigate the prevalence of Frailty in community older residents.
   * To explore the causes and risk factors of frailty.
2. Method:

   * The survey is a Community-based, multicenter prospective cohort study.

     1). 6,000 participants are expected to be included.
   * Through a questionnaire and physical examination form, carries on the investigation to the more than 65 years old people during the 3-year follow-up period.
   * The questionnaires include survey date, participant characteristics and related risk factors, such as comprise demographic characteristics, Chinese ethnic nationality, marital status, education level, family incomes, occupation, pregnancy and parity history, menstrual history, frequency and amount of daily smoking and alcohol drinking, frequency of urination and defecation, dietary habits, hours per day of sleep and sun exposure. Medical history including medication use and disease status for comorbidities, will be obtained from participants' medical records. Syndrome differentiation of deficiency of the five zang-organs in TCM will be analyzed.
   * Height and body weight will be measured for body mass index (BMI) calculation. The waist circumference and hip circumference will be recorded, and the ratios calculated. The muscle strengths of both hands will be measured with a hand dynamometer. Each of these measures will be assessed twice and the average score used in analyses.
   * Subjects will be asked to walk a distance of 4 meters and record the time at the same time to measure the walking speed.
   * Clock Drawing Test (CDT), physical frailty examination, Mini-Mental State Examination (MMSE), Skeletal muscle mass index (SMI) will also be conducted or calculated .
   * Each participant will provide a total of 7 mL of venous blood after an overnight fast (10-hour).

After being collected, markers of frailty will be measured, such as Interleukin-6 (IL-6), insulin-like growth factor-1 (IGF-1) and estrogen (E). And blood routine, urine routine, liver and kidney function, fasting plasma glucose, serum lipid will be detected.

* Physicians in each community as the backbone, Shanghai Geriatric Institute of Chinese Medicine is responsible for personnel training.
* Shanghai community health service centers are responsible for organization and coordination.

ELIGIBILITY:
Inclusion Criteria:

* more than 65 years old
* Permanent residence in Shanghai and long-term residence in the community implemented by this project (more than five years)
* Be willing to and be able to join in the study and signed Informed consent.

Exclusion Criteria:

* Excluding the patients whose physical function is affected by diseases or disabilities such as stroke, Parkinson's disease, tumor, fracture, etc.
* Excluding schizophrenia, depression, anxiety and other mental diseases and dependent on drug control.
* If they were unable to complete the study survey.
* Unwilling to join in the study and don't sign Informed consent.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Cluster random sampling was used in urban and rural areas of Shanghai
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The level of frailty | baseline
  1. Unexpected significant weight loss（>5%).
  2. Decreased strength: male grip strength ≤25 kg and female grip strength ≤18 kg
  3. Reduced physical activity in the last month.
  4. Slow walking speed is less than or equal to 0.8 m/s.
  5. How tired you feel for the last month? The frailty period was defined as ≥3 items, early frailty was defined as 1-2 items, and non-frailty was defined as 0 items.

SECONDARY OUTCOMES:
Clock Drawing Test | baseline
  The subjects were scored on a four-point scale by drawing a clock face on a piece of white paper.
Mini-Mental State Examination (MMSE) | baseline
  Two or three points in the drawing clock test were measured using the MMSE.
Skeletal muscle mass index (SMI) | baseline
  The ratio of skeletal muscle weight to height squared was measured by DXA.
Markers of frailty | baseline
  Markers of frailty, such as Interleukin-6 (IL-6), insulin-like growth factor-1 (IGF-1) and estrogen (E).
Routine inspection | baseline
  Fasting peripheral blood collected 4ml. blood routine, urine routine, liver and kidney function, fasting plasma glucose, serum lipid.

CONTACTS AND LOCATIONS:
Overall Officials: Chuan Chen, Principal Investigator — Shanghai Geriatric Institute of Chinese Medicine
Locations (1):
- Shanghai Geriatric Institute of Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No